CLINICAL TRIAL: NCT05270629
Title: Supermicrosurgical Lymphvenous Bypass Intervention for Lymphedema Treatment
Brief Title: Supermicrosurgical Lymphvenous Bypass Intervention for Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202101384B0
Record Dates: First submitted 2022-02-28; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Lymphedema of Leg

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lower limb lymphedema patients: This was a retrospective cohort propensity score-matched study. Patients with lower limb lymphedema were enrolled.
  Interventions: Other: Antegrade and retrograde anastomoses; Other: Antegrade-only anastomoses

INTERVENTIONS:
Other: Antegrade and retrograde anastomoses — Patients who had received both antegrade and retrograde anastomoses.
Other: Antegrade-only anastomoses — Patients who had received antegrade-only anastomoses.

SUMMARY:
Background: In addition to antegrade anastomosis, retrograde anastomosis has been thought to offer further improvements after lymphaticovenous anastomosis (LVA) by bypassing the retrograde lymphatic flow. However, this concept has yet to be validated. The aim of this study was to determine the impacts on outcomes of performing both retrograde and antegrade anastomosis, as compared to antegrade-only anastomosis for treating lower limb lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Lower limb lymphedema patients.

Exclusion Criteria:

* Patients who have had previous LVA, liposuction, or excisional therapy such as the Charles procedure were excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age > 18 years) with lower limb lymphedema patients were enrolled from March 2016 to December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-05 (Estimated)

PRIMARY OUTCOMES:
Magnetic resonance volumetry | 6 months after LVA
  Magnetic resonance volumetry was used for outcome assessments. The primary endpoint was the volume change at 6 months after LVA.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan